CLINICAL TRIAL: NCT04360785
Title: Effect of Two Methotrexate Injections in Sync With the First Adalimumab Injection to Prevent the Immunisation Anti Adalimumab During Treatment of Spondyloarthritis
Brief Title: Effect of Two Methotrexate in Sync With the First Adalimumab to Prevent the Immunisation Anti Ada in Spondyloarthritis
Acronym: MESYNAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP180571
Record Dates: First submitted 2020-03-02; First posted 2020-04-24 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-04

CONDITIONS: Spondyloarthritis
Keywords: adalimumab; anti-drug antibodies; tolerization; methotrexate; spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate + Adalimumab (Experimental): Experimental group : patients will receive 2 subcutaneous injections of methotrexate in addition of the usual adalimumab
  Interventions: Drug: Methotrexate
- Adalimumab (No Intervention): Reference group : patient will receive adalimumab as usual to treat spondyloarthritis

INTERVENTIONS:
Drug: Methotrexate — Patients randomized in this arm will have one subcutaneous injection of methotrexate 15min before and one 24h after their first injection of adalimumab prescribed as usual
  Arms: Methotrexate + Adalimumab

SUMMARY:
Preliminary report have demonstrated that methotrexate induces an anti bio-medicament tolerization whan administrated just before the first administration of the bio-medicament. Once this tolerization is obtained it seems useless to continue the methotrexate because this treatment has no efficacity in cases of spondyloarthritis.

DETAILED DESCRIPTION:
spondyloarthritis are treated in first intention by NSAIDs but in case of inefficacity biotherapies that inhib the TNF are used. Adalimumab is the most used anti TNF in this indication. Monoclonal antibody uses in therapy is immunogene, and there is a clear link between increase of anti drug antibody and in one hand decrease of drug serum concentration and in an other failure of the therapeutic response. With adalimumab there is an apparition of ADAb in 30%. There are reports suggesting that adding methotrexate to the therapy in a specific timeline allow to prevent the immunization. A previous study shows that association in long terms between methotrexate and adalimumab induce less immunized patients. The investigator's goal is to assess if two methotrexate subcutaneous injections at day 1 and 2 could prevent anti adalimumab antibodies formation.

ELIGIBILITY:
Inclusion criteria :

* Patients aged from 18 to 90
* Patients suffering from axial SpA, radiographic or non-radiographic according to ASAS criteria (peripheral involvement and/or Inflammatory bowel diseases could be present).
* Indication for anti TNF treatment: resistance to at least 2 NSAIDs and no contraindication to adalimumab
* No previous treatment with methotrexate in the last 3 months
* Stable dosage of steroids (less than 10mg/day of prednisone equivalent) and/or of NSAIDs for at least 10 days
* Contraception feminine or masculine
* Informed and written consent
* Social insurance

Exclusion criteria :

* Contraindication to methotrexate
* Previous treatment with adalimumab
* Steroids more than 10mg/day of prednisone equivalent
* Previous treatment with:

  * Etanercept in the last month
  * Infliximab, golimumab, certolizumab in the last 2 months (Previous treatment hereafter these dates with anti-TNF except adalimumab or secukinumab are not a counterindication)
* Current immunosuppressive drugs except methotrexate
* Current and proven pregnancy
* Project of pregnancy in the next 3 months following inclusion
* Legal safeguards
* Inclusion in another interventional research project

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
serum concentrations of ADAb anti adalimumab | 6 month
  To assess if 2 subcutaneous injections of methotrexate could prevent anti adalimumab antibodies formation at month 6 in patients with spondyloarthritis

SECONDARY OUTCOMES:
residual serum concentration of adalimumab | At 1, 3, 6 and 12 months
  To compare trough levels of adalimumab at month 1, 3, 6 and 12 in the 2 groups.
serum concentrations of ADAb anti adalimumab | At 1, 3 and 12 months
  To compare the percentage of immunized patients at month 1, 3 and 12 in the 2 groups
Incidence of Treatment-Emergent Adverse Events | At 1, 3, 6 and 12 months
  Incidence of Treatment-Emergent Adverse Events as assessed by the number of AE and SAE related to the treatment that occur during the participation of the patient
Comparison of Adalimumab Therapeutic efficacity in term of Activity disease using ASDAS (Ankylosing Spondylitis Disease Activity Score) score. | At 3, 6 and 12 months
  A therapeutic efficacity will be described as a clinical pertinent change of ASDAS : Ankylosing Spondylitis Disease Activity Score (at least 1,1 point) (a higher score means a worse outcome)
Comparison of Adalimumab Therapeutic efficacity in term of Activity disease using BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) score. | At 3, 6 and 12 months
  A therapeutic efficacity will be described as a clinical pertinent change of BASDAI : Bath Ankylosing Spondylitis Disease Activity Index (0 to 50 points - a higher score means a worse outcome)
Comparison of Adalimumab Therapeutic efficacity in term of therapeutic maintenance | At 3, 6 and 12 months
  Assess by Number of patient who didn't switch treatment
Comparison of Adalimumab Therapeutic efficacity in term of nonsteroidal anti inflammatory drugs ' reduction | At 3, 6 and 12 months
  Assess by ASAS-NSAIDS score (Assessment of SpondyloArthritis international Society - nonsteroidal antiinflammatory drugs) (minimum 0. a higher score means a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: gaetane Nocturne, Principal Investigator — APHP
Locations (17):
- France (17):
  - Hopital Pellegrin, Bordeaux
  - Hopital Ambroise Paré, Boulogne-Billancourt
  - Hopital La Cavale Blanche, Brest
  - CHU Trousseau, Chambray-lès-Tours
  - CH Sud Francilien, Corbeil-Essonnes
  - Hopital Mondor, Créteil
  - Kremlin Bicetre hospital, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - Hopital Saint Philibert, Lille
  - CHU Nantes, Nantes
  - CHR Orléans, Orléans
  - Hopital Bichat, Paris
  - Hopital Cochin, Paris
  - Hopital la Pitié Salpétrière, Paris
  - Hopital Saint Antoine, Paris
  - CH Pontoise, Pontoise
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No